CLINICAL TRIAL: NCT03541668
Title: A Phase III Trial to Assess the Efficacy and Safety of Recombinant Human Prourokinase in the Treatment of Acute Acute Ischaemic Stroke in 4.5 Hours After Stroke Onset
Brief Title: Study of rhPro-UK in Patients With Acute Ischaemic Stroke in 4.5 Hours After Stroke Onset(PROST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASLY-B1440-CTP-Ⅲa
Record Dates: First submitted 2018-03-13; First posted 2018-05-30 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2019-12

CONDITIONS: Acute Ischaemic Stroke
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Recombinant human urokinase (rhPro-UK)
  Interventions: Drug: Recombinant human urokinase
- Group B (Active Comparator): Alteplase(rt-PA)
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Recombinant human urokinase — Patients receive rhPro-UK 35mg,15mg of which is given as a bolus within 3 minutes followed by dlivery of the remaining 20 mg as a constant infusion over a period of 30 minutes.
  Other Names: rhPro-UK
  Arms: Group A
Drug: Alteplase — Patients receive rt-PA in a dose of 0.9mg per kilogram of body weight(maximum,90 mg),10 percent of which was given as a blous followed by delivery of the remaining 90 percent as a constant infusion over a period of 60 minutes.
  Other Names: rt-PA
  Arms: Group B

SUMMARY:
This is a randomized, rt-PA controlled, open-label phase 3 clinical study to evaluate the efficacy and safety of recombinant human urokinase(rhPro-UK) versus rt-PA thrombolysis for patients with acute ischaemic stroke in 4.5 hours after stroke onset.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke with symptoms of neurological deficits.
2. Aged 18 to 80 years（including the critical value）.
3. NIH Stroke Scale（NIHSS）scores of 4 to 25（including the critical value）.
4. Treatment within 4.5 hours after stroke onset.
5. The symptoms of stroke last at least 30 minutes without significant improvement before treatment.
6. CT showed negative or signs of early infarction.
7. Informed Consent Form signed by the patients or family (legal representatives) must be provided.

Exclusion Criteria:

1. Patients with premorbid modified Rankin Scale (mRS) score ≥2
2. CT showed multiple infarctions（low density> 1/3 cerebral hemisphere）.
3. Transient ischemic attack.
4. Epileptic seizure after stroke.
5. Intracranial tumor, arteriovenous malformation and aneurysm.
6. Iatrogenic Stroke.
7. Planned for thrombectomy.
8. Cardioembolism and atrial fibrillation.
9. Myocardial infarction history within 3 months.
10. Severe cerebral trauma or stroke history within 3 months.
11. Patients with systolic blood pressure ≥ 180mmHg or diastolic blood pressure ≥ 100mmHg after anti-hypertension treatment.
12. Intracranial hemorrhage or subarachnoid hemorrhage on baseline.
13. Active visceral hemorrhage.
14. Patients with intracerebral hemorrhage history.
15. Patients with diabetic retinopathy history.
16. Puncture in 1 week which can not be oppressed.
17. Major surgery or severe trauma within 2 weeks.
18. Intracranial surgery, intraspinal surgery or solid organ biopsy within 30 days.
19. Heparin treatment within 48h and increased APTT is above ULN.
20. Using of oral anticoagulant drugs and PT >15s or INR >1.7.
21. High risk of acute hemorrhage include platelet count<10^9/L.
22. Using of thrombin inhibitors or factor Xa inhibitor with abnormal results of sensitive laboratory examination.
23. Blood glucose < 2.7 mmol/L or > 22.2 mmol/L.
24. Pregnancy, lactating or menstrual women.
25. The investigator believes that the patient is not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-05-24 (Actual)

PRIMARY OUTCOMES:
Functional handicap | 90days
  Proportion of patients achieving a Modified Rankin Scale(mRS,which has a range of 0 to 6, with 0 indicating no symptoms at all and 6 indicating death) of 0 to 1 at 90 days after treatment.

SECONDARY OUTCOMES:
Proportion of Neurological Improvement | 90 days
  Proportion of patients achieving a NIHSS(national institutes of health stroke scale) ≦1 or reduction of ≥4 NIHSS points at 24 hours after treatment.
Scores of Neurological Improvement | 24 hours
  NIHSS changes from baseline at 24 hours after treatment
Long-term Change from Baseline | 90 days
  NIHSS, mRS and Barthel Index(which assesses the ability to perform activities of daily living, on a scale that ranges from 0 to 100) changes from baseline on 90 days after treatment.
Proportion of Long-term Improvement | 90 days
  Proportion of patients achieving a mRS of 0 to 2 and a Barthel Index of 75 to 100 at 90 days after treatment.
Systemic hemorrhage | 90days
  Severe systemic hemorrhage
Symptomatic intracerebral hemorrhage | 90days
  Symptomatic intracerebral hemorrhage (sICH)
Death | 7 days and 90 days
  Death
Recurrence | 7 days
  Recurrence of stroke
Liver function | 7 days
  The incidence of ALT≥3ULN in liver biochemical examination
Renal function | 7 days
  The incidence of Scr rising to 3 times or ≥ 4mg/dl more than the base value

CONTACTS AND LOCATIONS:
Locations (35):
- China (35):
  - Beijing Luhe Hospital,Capital Medical University, Beijing, Beijing Municipality
  - XuanWu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The First Hospital of Handan, Handan, Hebei
  - Harrison International Peace Hospital, Hengshui, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Changsha, Changsha, Hunan
  - First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - The Second People'Hospital of Huai'an, Huai'an, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - The Neuropsychiatric Hospital of Jilin Province, Siping, Jilin
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Shenyang Military Region General Hospital, Shenyang, Liaoning
  - The 163th Hospital of the Chinese People's Liberation Army, Shenyang, Liaoning
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The People's Hospital of Sichuan Province, Chengdu, Sichuan
  - Deyang people's hospital, Deyang, Sichuan
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Luoyang Central Hospital, Luoyang, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song H, Wang Y, Ma Q, Feng W, Liu R, Lv X, Huang L, Li Y, Yang Y, Geng D, Zhu J, Wei Y, Chen H, Zhu R, Zhai Q, Guo J, Liu B, Zhao S, Wang Y; PROST collaborative group. Efficacy and Safety of Recombinant Human Prourokinase in the Treatment of Acute Ischemic Stroke Within 4.5 Hours of Stroke Onset: A Phase 3 Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2325415. doi: 10.1001/jamanetworkopen.2023.25415. PMID 37490291